CLINICAL TRIAL: NCT06266663
Title: Social Determinants of Health, Medication Use, and Quality of Life in Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-13788; CNTO1275IBD4012 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — A cross-sectional survey of 400 IBD patients who will be actively recruited from the gastroenterology (GI) specialty clinics at Einstein-Montefiore Medical Center and Icahn School of Medicine at Mount Sinai Hospital. The survey will consist of validated screening measures on social domains known to affect health outcomes as well as measures of medication adherence and HRQoL.

SUMMARY:
Optimizing health related-quality of life (HRQoL) for patients with inflammatory bowel disease (IBD), who often experience a relapsing disease course, is an essential component of care. Improving IBD disease control is linked to increased health-related quality of life. Even as many effective pharmacotherapies to promote disease control are available, evidence suggests that Hispanic and Non-Hispanic Black IBD patients may not receive full benefit from these therapies compared to their Non-Hispanic White counterparts. Underlying mechanisms that contribute to observed disparities in the use of IBD medical therapies are likely multifactorial. Adequate access to treatment has been implicated. Hispanic and Non-Hispanic Black IBD patients are more likely to be Medicaid-insured, and Medicaid insurance has been associated with increased emergency room visits, a proxy for sub-optimal IBD control. Medication adherence has also been proposed as a potential mediating factor. IBD therapies can be time-consuming and costly, which can pose a challenge in achieving medication adherence. While previous studies suggest Black IBD patients have lower medication adherence than Non-Hispanic White patients, it is unclear the extent to which social factors contribute to this observation. The purpose of this study is to evaluate the association between social determinants of health, medication adherence, and HRQoL among Hispanic and Non-Hispanic Black IBD patients. Understanding potentially modifiable psychosocial factors that contribute to medication adherence and HRQoL will provide targets for later intervention towards the goal of health equity.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Crohn's disease, ulcerative colitis, or indeterminate colitis ≥ 3 months investigator confirmed on the basis of supportive clinical data such as colonoscopy, pathology and/or radiology
* age 18 years or older
* ability to provide informed consent in English or Spanish
* basic computer proficiency (i.e. to complete online survey)

Exclusion Criteria:

* race and ethnicity self-identified as other than Hispanic, Non-Hispanic Black, or Non-Hispanic White

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients age 18 years or older with IBD who meet the above inclusion/exclusion criteria will be eligible to participate in the study. Participants will be grouped by race and ethnicity (Hispanic, Non-Hispanic Black, or Non-Hispanic White). Participants who identify as Hispanic will be further grouped by preferred language (English or Spanish). Participants will also be grouped into either public (e.g. Medicaid, Medicare) or private insurance. The study team plans to recruit 25 participants per cell: race and ethnicity (4), study site (2), insurance (2). Target recruitment is 200 participants per site for a total of 400 participants.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
IBD medication adherence | Single 20 minute survey response, upon participant enrollment
  The outcome of IBD medication adherence will be categorized by the adapted Hill Bone Medication Adherence Scale (HB-MAS). This part of the questionnaire consists of eight items used to assess patients' self-reported IBD oral medication adherence. Participant responses are scored on a scale from 1-4 (1 = All of the time; 2 = Most of the time; 3 = Some of the time; 4 = None of the time). Lower overall scores are associated with better medication adherence
Health-related quality of life (HRQoL) | Single 20 minute survey response, upon participant enrollment
  HRQoL will be categorized based on responses to the NIH Patient Reported Outcomes Measurement Information System-29 (PROMIS-29). PROMIS-29 assesses each of 7 domains (Depression, Anxiety, Physical function, Pain interference, Fatigue, Sleep disturbance, Ability to participate in social roles and activities) using 4 questions with an additional Pain Intensity question. Participants' responses are scored from 1-5 (with the exception of the Pain Intensity Question which is scored from 0-10). The sum of each of the 7 PROMIS domains results in a raw score (from 4-20). There is no total score. Each axis forms its own score. PROMIS assessments use an Item Response Theory (IRT) based score called "Expected A Posteriori" or EAP scores, which are then transformed to a final T-score metric. As such, scores are mapped so that the values follow a normal distribution with a population mean T-score of 50 and a standard deviation of 10

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Greywoode, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Hutchinson Campus, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szigethy EM, Allen JI, Reiss M, Cohen W, Perera LP, Brillstein L, Cross RK, Schwartz DA, Kosinski LR, Colton JB, LaRusso E, Atreja A, Regueiro MD. White Paper AGA: The Impact of Mental and Psychosocial Factors on the Care of Patients With Inflammatory Bowel Disease. Clin Gastroenterol Hepatol. 2017 Jul;15(7):986-997. doi: 10.1016/j.cgh.2017.02.037. Epub 2017 Mar 12. PMID 28300693
- [Background] Kappelman MD, Long MD, Martin C, DeWalt DA, Kinneer PM, Chen W, Lewis JD, Sandler RS. Evaluation of the patient-reported outcomes measurement information system in a large cohort of patients with inflammatory bowel diseases. Clin Gastroenterol Hepatol. 2014 Aug;12(8):1315-23.e2. doi: 10.1016/j.cgh.2013.10.019. Epub 2013 Oct 29. PMID 24183956
- [Background] Nguyen GC, LaVeist TA, Harris ML, Wang MH, Datta LW, Brant SR. Racial disparities in utilization of specialist care and medications in inflammatory bowel disease. Am J Gastroenterol. 2010 Oct;105(10):2202-8. doi: 10.1038/ajg.2010.202. Epub 2010 May 18. PMID 20485281
- [Background] Damas OM, Jahann DA, Reznik R, McCauley JL, Tamariz L, Deshpande AR, Abreu MT, Sussman DA. Phenotypic manifestations of inflammatory bowel disease differ between Hispanics and non-Hispanic whites: results of a large cohort study. Am J Gastroenterol. 2013 Feb;108(2):231-9. doi: 10.1038/ajg.2012.393. Epub 2012 Dec 18. PMID 23247580
- [Background] Barnes EL, Loftus EV Jr, Kappelman MD. Effects of Race and Ethnicity on Diagnosis and Management of Inflammatory Bowel Diseases. Gastroenterology. 2021 Feb;160(3):677-689. doi: 10.1053/j.gastro.2020.08.064. Epub 2020 Oct 21. PMID 33098884
- [Background] Nguyen GC, Sam J, Murthy SK, Kaplan GG, Tinmouth JM, LaVeist TA. Hospitalizations for inflammatory bowel disease: profile of the uninsured in the United States. Inflamm Bowel Dis. 2009 May;15(5):726-33. doi: 10.1002/ibd.20825. PMID 19067416
- [Background] Nguyen GC, LaVeist TA, Harris ML, Datta LW, Bayless TM, Brant SR. Patient trust-in-physician and race are predictors of adherence to medical management in inflammatory bowel disease. Inflamm Bowel Dis. 2009 Aug;15(8):1233-9. doi: 10.1002/ibd.20883. PMID 19177509